CLINICAL TRIAL: NCT05796583
Title: Pulsed Electromagnetic Fields for Postoperative and Post-Amputation Analgesia: A Randomized, Participant- and Observer-Masked, Sham-Controlled Pilot Study
Brief Title: Pulsed Shortwave Therapy for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSWT SofPulse
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment: Randomized, Triple-Masked, Placebo-Controlled, Parallel-Arm Human Subjects Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Investigational Drug Service will create the randomization tables and provide the investigators with the appropriate device (active or sham), leaving all participants, investigators, and the statistician masked to treatment group assignment with the exception of the study coordinator who receives the study device from the Investigational Drug Service.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Pulsed Shortwave Treatment with SofPulse (Active Comparator): Application of 8 days of nonthermal, pulsed shortwave (radiofrequency) therapy with Endonovo Therapeutics SofPulse
  Interventions: Device: Active Pulsed Shortwave Treatment
- Sham Treatment (Sham Comparator): Application of 8 days of sham device
  Interventions: Device: Sham Treatment

INTERVENTIONS:
Device: Active Pulsed Shortwave Treatment — Application of 8 days of nonthermal, pulsed shortwave (radiofrequency) therapy with Endonovo Therapeutics SofPulse
  Other Names: non thermal, pulsed shortwave (radio frequency) therapy; pulsed electromagnetic fields therapy
  Arms: Active Pulsed Shortwave Treatment with SofPulse
Device: Sham Treatment — Application of 8 days of a nonfunctional sham device
  Other Names: Placebo treatment
  Arms: Sham Treatment

SUMMARY:
Pulsed shortwave (radiofrequency) therapy is a possible method of pain control involving the application of electromagnetic energy (also termed pulsed electromagnetic fields). Food and Drug Administration-cleared devices have been in clinical use for over 70 years. For decades, available devices consisted of a large signal generator and bulky coil applicator that were not portable and produced significant electromagnetic interference, making them impractical for common use. However, small, lightweight, relatively inexpensive, noninvasive, Food and Drug Administration-cleared devices that function for 8 days are now available to treat acute and chronic pain, decrease inflammation and edema, and hasten wound healing and bone regeneration. Therefore, it has the potential to concurrently improve analgesia and decrease or even negate opioid requirements, only without the limitations of opioids and peripheral nerve blocks. The purpose of this study is to explore the possibility of treating acute postoperative pain with nonthermal, pulsed shortwave (radiofrequency) therapy, optimize the study protocol, and estimate the treatment effect.

DETAILED DESCRIPTION:
The proposed study will be a randomized, participant- and observer-masked, sham-controlled, parallel-arm, human participants study with two primary aims:

Specific Aim 1: To determine the feasibility and optimize the protocol for subsequent clinical trials that will compare the addition of nonthermal, pulsed shortwave therapy to usual and customary analgesia following moderate-to-severely painful surgical procedures.

Specific Aim 2: To estimate the treatment effect of adding nonthermal, pulsed shortwave therapy to usual and customary analgesia on pain and opioid consumption following moderate-to-severely painful surgical procedures.

Hypothesis 1 (primary): Nonthermal, pulsed shortwave therapy decreases pain in the 7 days following moderate-to-severely painful surgical procedures.

Hypothesis 2: Nonthermal, pulsed shortwave therapy decreases opioid use in the 7 days following moderate-to-severely painful surgical procedures.

This will be a single-center (University of California San Diego), randomized, participant- and observer-masked, sham-controlled, parallel-arm human subjects study.

Enrollment. Participants will be consenting adults undergoing various surgical procedures usually resulting in moderate-to-severe postoperative pain. Study inclusion will be proposed to eligible presurgical patients. If an individual desires study participation, written, informed consent will be obtained using a current University of California San Diego Institutional Review Board-approved informed consent form. The study population of interest includes adult women and men of all races, ethnicity, sexual identity, and socioeconomic status.

Procedures. Following written, informed consent, we will record baseline anthropometric information (age, sex, height, weight, amputation details and current pain levels). Participants will receive any standard peripheral nerve block(s) administered using bupivacaine or ropivacaine 0.5% with epinephrine (standard at University of California San Diego) prior to undergoing their surgical procedure per standard of care.

Treatment Group Assignment. Each participant will be randomized to one of two treatment groups: Active or Sham treatment. Randomization will be stratified by surgical procedure in block sizes of 2. The computer-generated randomization lists will be created by the University of California San Diego Investigational Drug Service in a 1:1 treatment group ratio. An Investigational Drug Service pharmacist will provide the investigators with the appropriate device. Upon completion of data collection for a specific subgroup (e.g., total knee and hip arthroplasty; cholecystectomy), the pharmacist will provide the investigators with a masked list of the treatment groups (e.g., "Treatment A" and "Treatment B"), and the active/sham lists only following analysis for that subgroup, resulting in a triple-masked study (investigators, participants, statistician).

Study intervention. The pulsed shortwave device will be affixed over the primary wound area(s) using tape and activated prior to recovery room discharge. The optimal location to treat phantom pain is currently unknown and will partially informed by the results of this study, and patients will be encouraged to move the devices to a new anatomic location until relief is optimized.

Supplemental analgesics. In addition to the pulsed shortwave device, participants will receive standard-of-care supplemental analgesics. Therefore, all patients of this study-regardless of the treatment arm they are randomized to-will continue to receive current usual and customary analgesia: all will receive the same combination of supplemental analgesics they would regardless of study participation. Participants (and their caretakers) will be provided with verbal and written instructions, and the telephone and pager numbers of an investigator available during business hours throughout the treatment period. Participants cannot shower or submerge the device, as advised by the manufacturer; but will be allowed to remove it to bathe, and subsequently replace the device following bathing.

Participants will be discharged with their pulsed shortwave device in situ and a prescription for immediate-release oral opioid, preferably oxycodone 5 mg tablets, taken for breakthrough pain (surgeons occasionally prefer a different type of opioids such as hydrocodone, which is why we analyze the data using oral oxycodone equivalents). The pulsed shortwave devices will be removed by participants at home following Day 8 when the battery is exhausted. Removing the devices encompasses tape removal and discarding (these are disposable, single-use devices).

Outcome measurements (end points). We have selected outcome measures that have established reliability and validity, with minimal inter-rater discordance, and are recommended for pain-related clinical trials by the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consensus statement. All data collection will be through standard UCSD EPIC notes and patient interviews in-person during hospitalization or via a telephone call for outpatients. Postoperatively, surgical endpoints will be recorded such as surgical duration. All pain scores will be measured using the Numeric Rating Scale (0: no pain, 10: worst imaginable pain).

Statistical plan and sample size estimation. there will be a total of 70 surgical participants, and these patients will be analyzed separately from Phase I surgical and amputation patients. Sample size calculations are based upon the hypothesis that pulsed electromagnetic field therapy decreases pain in the 7 days following moderate-to-severely painful surgical procedures. The primary outcome calculated as follows: for each participant all of the "average" and "worst" daily pain scores collected within the first 7 postoperative days will be summed. We will use these summed scores from participants having cholecystectomy (n=30), and hip and knee arthroplasty (n=40) to estimate a probable sample size.

We will consider a 33% reduction in pain scores to be the minimal clinically important difference [Farrar et al. J Pain Symptom Management 2003; 25: 406-11]. Based on values from patients receiving sham in an (as-of-yet) unpublished pilot study, we anticipate the sham group to have an anticipated mean (SD) of 23.9 (12.3). Assuming a two-sided type I error protection of 0.05 and a power of 0.80, approximately 25 patients in each group are required (ClinCalc.com, accessed 2/23/23). To allow for a higher degree of variability than anticipated we will enroll a total of 70 participants: cholecystectomy (n=30), and hip and knee arthroplasty (n=40).

Continuous, normally-distributed data will be reported as mean ± standard deviation. Nonparametric continuous or categorical data will be reported as median [10th-90th percentiles] or precents, as appropriate. Comparisons of independent samples will be performed using Student's t-test for parametric continuous variables or Mann-Whitney U test for nonparametric or categorical variables. The Chi Square test and Fisher's Exact test will be used for differences in proportions, as appropriate. P<0.05 will be considered statistically significant for the primary outcome. Results of comparisons in secondary outcomes will be interpreted as suggestive, requiring confirmation in a future trial before considering them as definitive.

ELIGIBILITY:
Adult patients of at least 18 years of age undergoing one of these primary surgical procedures:

* primary knee arthroplasty
* primary hip arthroplasty
* cholecystectomy

Exclusion Criteria:

* concurrent use of an implanted pulse generator (e.g., cardiac pacemaker)
* pregnancy
* incarceration
* chronic opioid/tramadol use (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
* neuro-muscular deficit of the surgical area/limb
* a planned postoperative perineural local anesthetic infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ilfeld BM, Finneran JJ 4th, Said ET, Ball ST, Sandler BJ, Broderick RC, Gonzales FB, Lau NJ, Schaar A, Abdullah B. Pulsed Shortwave (Radiofrequency) Therapy With a Noninvasive, Wearable, Disposable Device: A Randomized, Participant- and Assessor-Masked, Sham-Controlled Pilot Study. Neuromodulation. 2025 Jun;28(4):682-689. doi: 10.1016/j.neurom.2025.01.008. Epub 2025 Feb 20. PMID 39985539

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (16) | 58 (17) | 55 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 9 | 11 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Height [Mean (Standard Deviation); unit: cm] | 165 (10) | 168 (10) | 166 (10)
Weight [Mean (Standard Deviation); unit: kg] | 81 (30) | 87 (23) | 84 (26)

OUTCOME MEASURES:

1. Primary Outcome: Pain Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. The primary outcome calculated as follows: for each participant all of the "average" and "worst" daily pain scores collected within the first 7 postoperative days will be summed: specifically on Days 1, 2, 3, and 7, resulting in a scale of 0-80.
Time Frame: First postoperative week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 28 (11) | 34 (14)

2. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 3.4 (2.1) | 3.8 (2.3)

3. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 2.4 (1.9) | 3.3 (2.0)

4. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 2.1 (1.9) | 3.4 (1.9)

5. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 1.0 (1.3) | 2.2 (1.8)

6. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | .9 (1.6) | 1.4 (1.9)

7. Secondary Outcome: AVERAGE Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | .2 (1.2) | .3 (1)

8. Secondary Outcome: Median AVERAGE Pain Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. The outcome will the mean value of daily average pain scores measured with the Numeric Rating Scale.
Time Frame: Median value of the average daily pain measured on postoperative days 1, 2, 3, and 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 1.8 [0.5 to 3.4] | 3.3 [1.9 to 4.3]

9. Secondary Outcome: Median WORST Pain Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. The outcome will the median value of daily worst pain scores measured with the Numeric Rating Scale.
Time Frame: Median value of the worst daily pain measured on postoperative days 1, 2, 3, and 7
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 5.0 [4 to 5.9] | 5.5 [3.6 to 7.1]

10. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 6.3 (2) | 6.8 (2.4)

11. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 5.3 (2.5) | 5.9 (2.2)

12. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 4.7 (2.3) | 5.1 (2.6)

13. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 2.7 (1.7) | 4 (2.5)

14. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | 2.3 (2.1) | 2.8 (2.6)

15. Secondary Outcome: WORST Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | .3 (1.6) | .6 (1.6)

16. Secondary Outcome: LEAST Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | .4 (.9) | .9 (1.5)

17. Secondary Outcome: LEAST Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | .3 (.8) | .4 (1.3)

18. Secondary Outcome: CURRENT Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | .8 (1.2) | 1.6 (1.2)

19. Secondary Outcome: CURRENT Pain Measured With the Numeric Rating Scale
Description: as for outcome 2
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
units on a scale | .6 (1.2) | 1.2 (1.9)

20. Secondary Outcome: Total OPIOID Consumption for Postoperative Days 1, 2, 3, and 7 (Measured in Oral Oxycodone Equivalents)
Description: Cumulative opioid consumption queried on postoperative days 1, 2, 3, and 7 (measured in oral oxycodone equivalents).
Time Frame: Cumulative opioid consumption queried on postoperative days 1, 2, 3, and 7
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
mg | 4.6 (4.9) | 5.1 (7.3)

21. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
mg | 2.1 (2.4) | 2 (3.2)

22. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
mg | 1.6 (2.2) | 1.4 (2.7)

23. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
mg | .7 (1.1) | 1.2 (2.3)

24. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
mg | .3 (.9) | .9 (1.7)

25. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
mg | .4 (1) | .6 (1.9)

26. Secondary Outcome: Opioid Consumption of the Previous 24 Hours (Measured in Oral Oxycodone Equivalents)
Description: Opioid consumption of the previous 24 hours (measured in oral oxycodone equivalents)
Time Frame: postoperative day 180
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
mg | 0.1 (.6) | .0 (0)

27. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Subscale)
Description: The Brief pain Inventory short form interference sub scale is an instrument specifically designed to assess pain and its impact on physical and emotional functioning which includes 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference;10=complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. The final scale is from 0 (no interference) to 70 (maximum interference).
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
score on a scale | 9.3 (12.4) | 12 (13.6)

28. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Subscale)
Description: as for outcome 27
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
score on a scale | 6.5 (12.6) | 9 (13)

29. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
number of awakenings | .7 (1.3) | 1.1 (2.2)

30. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 2
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
number of awakenings | .4 (.8) | .7 (1.2)

31. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
number of awakenings | .3 (.9) | 1.1 (2)

32. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 7
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
number of awakenings | .5 (1.1) | .5 (1.2)

33. Secondary Outcome: Awakenings Due to Pain
Description: The number of times the participant awoke the previous night due to pain
Time Frame: postoperative day 14
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
number of awakenings | .3 (.8) | .9 (2)

34. Secondary Outcome: Hospitalization Duration Measured in Days
Description: Day relative to the day of surgery that patient was discharged from the hospital (e.g., same day is postoperative day 0, while the day following surgery is postoperative day 1)
Time Frame: First postoperative week
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
Days | .4 (.7) | .4 (.7)

35. Secondary Outcome: Surgical Duration
Description: The time from surgical start to surgical stop measured in minutes
Time Frame: intraoperative (within the operating room)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
minutes | 78 (27) | 88 (33)

36. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one or both of the intervention devices (and where the device is moved to) since the last phone contact
Time Frame: postoperative day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

37. Secondary Outcome: Device Location Changes
Description: as for outcome 36
Time Frame: postoperative day 2
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

38. Secondary Outcome: Device Location Changes
Description: as for outcome 36
Time Frame: postoperative day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

39. Secondary Outcome: Device Location Changes
Description: as for outcome 36
Time Frame: postoperative day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

40. Secondary Outcome: Device Location Changes
Description: as for outcome 36
Time Frame: postoperative day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

41. Secondary Outcome: Passive Joint Flexion
Description: The number of degrees the patient can flex their knee or hip (for these procedures only; cholecystectomy excluded)
Time Frame: postoperative day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
Number analyzed (Participants) | 35 | 35
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months following surgery
Arm/Group | Active Pulsed Shortwave Treatment With SofPulse | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT05796583/Prot_SAP_000.pdf